CLINICAL TRIAL: NCT02571166
Title: Phase I Study of the Genital Immune Response to Live, Attenuated HSV529 Vaccine in HSV-2 Seropositive Adults
Brief Title: HSV529 Vaccine in HSV-2 Seropositive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49596-J; 8377 (Other: Fred Hutch/UW Cancer Consortium IRB)
Record Dates: First submitted 2015-08-13; First posted 2015-10-08 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Herpes Simplex Virus 2
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSV529 (Experimental)
  Interventions: Biological: HSV529; Drug: Valacyclovir

INTERVENTIONS:
Biological: HSV529 — Live, Replication-defective HSV-2 virus
Drug: Valacyclovir — 500 mg orally, once daily for 4 weeks

SUMMARY:
The purpose of the study is to determine the safety of HSV529 vaccine in healthy volunteers with HSV infection and to determine if administration of the HSV529 vaccine increases the immune response in genital skin.

DETAILED DESCRIPTION:
The investigators will enroll a cohort of 8-10 HIV-1 seronegative, HSV-2 seropositive persons with recurrent genital HSV-2 lesions in an area amenable to genital biopsy. Participants will enroll when they have a genital lesion. They will undergo a lesion biopsy and a non-lesion biopsy. They will start suppressive valacyclovir 500 mg po daily for 4 weeks. Three days after completion of the 4 week valacyclovir course, participants will initiate vaccination with HSV529 on a 0, 1, and 6 month dose schedule. At each vaccination visits and at the 10 days post vaccination visits, genital biopsies will be performed. Genital biopsies will be performed at the site of genital lesion and at a non-lesional genital site. PBMC will also be drawn. Two days after the second vaccination, an optional biopsy will be offered. Overall, a minimum of 14 genital biopsies will be performed for each participant: 7 at the genital lesion site, and 7 at the genital non-lesion site. Four control biopsies from the upper arm will also be performed. For participants who undergo the optional biopsy two days after Dose 2, two additional genital biopsies will be performed. Participants will also collect daily genital swabs for HSV PCR for 30 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. HSV-2 seropositive by UW Western blot with a history of recurrent genital herpes, with lesions in an area amenable to biopsy.
2. Aged 18 to 55 years on the day of enrollment.
3. In good general health with absence of significant health problems as determined by medical history, physical examination, and laboratory screening performed during screening visits.
4. Hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, and liver function (ALT, AST, alkaline phosphatase, total bilirubin) screening laboratory results do not fall into the range of values that are Grade 1 or greater as per the toxicity grading scale.
5. Female subjects must be of non-childbearing potential i.e. surgically sterilized (bilateral tubal ligation, hysterectomy) or, if of child-bearing potential and sexually active with a male partner, she must be willing to use a highly effective method of contraception (e.g., intrauterine device (IUD); oral contraceptives, diaphragm or condom in combination with contraceptive foam, jelly or cream; Norplant, DepoProvera, contraceptive skin patch or cervical ring) for at least 30 days prior to vaccination and until 30 days after final vaccination or be in a monogamous relationship with a male partner who has undergone a vasectomy at least 6 months prior to first dose of HSV529.
6. Willingness to attend all scheduled visits and able to comply with all trial procedures (e.g., blood draws, biopsies, completion of diary cards, return for follow-up visits, accessible by phone or pager, able to self-sample for assessment of asymptomatic shedding of HSV, and not planning on moving from study area).
7. HIV seronegative.
8. Subject is willing not to use antiviral therapy 3 days before each injection and during swabbing periods. If recurrences occur during swabbing periods, participants will be asked NOT to take antiviral therapy.
9. Subject is willing to forgo receipt of a licensed, live vaccine in the 30 days preceding each dose of vaccine or in the 30 days following each dose of vaccine. The inactivated flu vaccine can be used ≥14 days before or ≥14 days after administration of study vaccine, if this is felt to be necessary.
10. Persons who have close contact with infants or immunocompromised individuals are willing to avoid such contact for 3 days after each injection.

Exclusion Criteria:

1. Subject is pregnant or nursing OR planning to become pregnant in the timeframe that begins 30 days prior to the first vaccination and ends 30 days after the third vaccination.
2. Body Mass Index greater than 35.
3. Hepatitis C seropositive
4. Hepatitis B surface antigen positive
5. Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination or planned participation during the study period up to 6 months after the last dose of vaccine. The non-interventional follow-up for an earlier study (e.g., long-term surveillance) will be allowed.
6. Severe active infection or serious HSV-2 related or unrelated medical conditions that, in the opinion of the investigator, would prevent study completion.
7. Subjects with 9 or more symptomatic recurrences of genital herpes disease within the year prior to Day 0.
8. A history of HSV infection of the eye (e.g., herpes simplex interstitial keratitis or uveitis).
9. A history of herpes gladiatorum, herpetic whitlow or eczema herpeticum.
10. A history of lesions caused by HSV on either arm.
11. A history of herpes-associated erythema multiforme.
12. A history of a clinically significant autoimmune disorder.
13. Known or suspected congenital or acquired immunodeficiency.
14. Receipt of anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
15. Subjects using corticosteroids (excluding topical, inhaled or nasal) or any immunomodulating drugs (see Prohibited Medications Section) within 42 days prior to the first vaccination. An immunosuppressive dose of corticosteroids is defined as ≥10 mg prednisone equivalent per day for >14 days.
16. Subjects without a spleen.
17. Subjects receiving immunoglobulin within the past 6 months or anticipated receipt of immunoglobulin during the 28 days following each vaccination.
18. Bleeding disorder, or receipt of anticoagulants that, in the opinion of the Investigator, would interfere with the subject's participation in the trial.
19. Known allergy or intolerance to vaccine components [e.g., potassium glutamate (possible cross-reaction to monosodium glutamate), sucrose] or to a vaccine containing any of the same substances.
20. Known allergy or intolerance to silver nitrate or lidocaine.
21. Known allergy or intolerance to acyclovir or valacyclovir.
22. Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
23. History of keloid formation or excessive scarring.
24. History of frequent cellulitis or boils (>3 episodes in past 2 years) requiring antibiotic therapy.
25. Prior receipt of an HSV vaccine.
26. Any condition that the PI thinks might compromise the person's ability to comply with the requirements of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Safety of HSV529 vaccine assessed by solicited Adverse Events, non-solicited Adverse Events and all Serious Adverse Events. | one year
  To determine the safety of HSV529 vaccine we will assess solicited Adverse Events, non-solicited Adverse Events and all Serious Adverse Events.
T cell density | one year
  Change in density of total CD4+, CD4+ Foxp3+, and CD8+ T cells in the genital mucosa at sites of lesions prior to and post HSV529 vaccination
TCR composition | one year
  Change in the diversity and clonality of TCR composition pre and post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, MPH, Principal Investigator — University of Washington; Lawrence Corey, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States